CLINICAL TRIAL: NCT01850017
Title: Prospective Randomized Double Blind Study of Intraoperative Dexmedetomidine and Postoperative Pain Control in Patients Undergoing Multi-level Thoraco-lumbar Spine Surgery
Brief Title: Study of Dexmedetomidine in Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bhiken I. Naik, MD, Assistant Professor, Anesthesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16150
Record Dates: First submitted 2013-04-30; First posted 2013-05-09 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Collapse of Thoracic Vertebra; Collapse of Lumbar Vertebrae
Keywords: Opiate consumption; Visual Analogue Scale
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone and dexmedetomidine (Experimental): Standard American Society of Anesthesiology monitors. Midazolam 1-2 mg for pre-operative sedation. Lidocaine 0.5-1 mg/kg with induction. Propofol 1-2 mg/kg with induction. Fentanyl 0.5-1 mcg/kg with induction. Rocuronium 0.5 -1 mg/kg with induction. Total intravenous anesthesia with propofol for maintainence of anesthesia. Titrated to maintain BIS (bispectral index) between 30-60.
  Methadone 0.2 mg/kg ideal body weight and dexmedetomidine 1 mcg/kg load over 20 minutes followed by a continuous infusion of 0.5 mcg/kg/h for the duration of the procedure.
  Interventions: Drug: Dexmedetomidine
- Methadone and placebo (No Intervention): Standard American Society of Anesthesiology monitors. Midazolam 1-2 mg for pre-operative sedation. Lidocaine 0.5-1 mg/kg with induction. Propofol 1-2 mg/kg with induction. Fentanyl 0.5-1 mcg/kg with induction. Rocuronium 0.5 -1 mg/kg with induction. Total intravenous anesthesia with propofol for maintainence of anesthesia. Titrated to maintain BIS (bispectral index) between 30-60.
  Methadone 0.2 mg/kg ideal body weight and placebo (normal saline) 1 mcg/kg load over 20 minutes followed by a continuous infusion of 0.5 mcg/kg/h for the duration of the procedure

INTERVENTIONS:
Drug: Dexmedetomidine — In the intervention arm dexmedetomidine at a dose of 1 mcg/kg over 20 mins followed by an infusion of 0.5 mcg/kg/h for the duration of the surgery.
  Other Names: Precedex
  Arms: Methadone and dexmedetomidine

SUMMARY:
The investigators will conduct a prospective randomized double blind study comparing methadone plus methadone and intraoperative dexmedetomidine in multi-level spine surgery in two randomized groups. The investigators plan to document the intraoperative opioid requirements, time to first dose of opioids postoperatively and total opioid consumption in the first 24, 48 and 72 hours. The incidence of intra and postoperative complications will be assessed.

DETAILED DESCRIPTION:
Patients presenting for thoracic and/or lumbar spine surgery with neuromonitoring (MEP/SSEP/EMG)will be recruited. Standard anesthesia monitoring will be performed. Randomized to a placebo or dexmedetomidine arm. Both groups will receive methadone 0.2 mg/kg ideal weight after induction of anesthesia.

The placebo/dexmedetomidine will be loaded at 1 mcg/kg over 20 minutes and then a continuous infusion of 0.5 mcg/kg/h for the duration of the procedure.

Intraoperative analgesia will be provided with fentanyl and dilaudid per the anesthesia team.

Upon closure the study drug will be terminated. Patients will be followed up for 72 hours after surgery. Total opiate consumption and visual analogue scale ratings will be documented.

Intra and postoperative inotrope/pressor requirements will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years of age
* Elective multi-level thoracic and/or lumbar spine surgery requiring SSEP, EMG or MEP monitoring

Exclusion Criteria:

* Emergency spine surgery
* Age < 18 years
* Pregnant patients
* Advanced heart block: Mobitz type II block or atrio-ventricular dissociation in a previous EKG.
* Any individual with stage 4 or greater chronic kidney disease (eGFR< 30 ml/min) and/or requiring dialysis or liver failure defined as a history of cirrhosis or fulminant hepatic failure
* Any individuals on preoperative methadone therapy
* Preoperative dexmedetomidine use
* Preoperative systolic hypertension defined by a systolic blood pressure greater than 150 mmHg in the surgical admission suite
* Enrolled in another study within 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Opiate consumption | 72 hours post surgery
  We will measure total opiate consumption 72 hours post surgery

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 72 hours
  We will measure pain scores on the Visual analogue scale after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bhiken Naik, MBBCh, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Korkmaz Dilmen O, Tunali Y, Cakmakkaya OS, Yentur E, Tutuncu AC, Tureci E, Bahar M. Efficacy of intravenous paracetamol, metamizol and lornoxicam on postoperative pain and morphine consumption after lumbar disc surgery. Eur J Anaesthesiol. 2010 May;27(5):428-32. doi: 10.1097/EJA.0b013e32833731a4. PMID 20173643
- [Background] Khan ZH, Rahimi M, Makarem J, Khan RH. Optimal dose of pre-incision/post-incision gabapentin for pain relief following lumbar laminectomy: a randomized study. Acta Anaesthesiol Scand. 2011 Mar;55(3):306-12. doi: 10.1111/j.1399-6576.2010.02377.x. PMID 21288211
- [Background] Loftus RW, Yeager MP, Clark JA, Brown JR, Abdu WA, Sengupta DK, Beach ML. Intraoperative ketamine reduces perioperative opiate consumption in opiate-dependent patients with chronic back pain undergoing back surgery. Anesthesiology. 2010 Sep;113(3):639-46. doi: 10.1097/ALN.0b013e3181e90914. PMID 20693876
- [Background] Grewal A. Dexmedetomidine: New avenues. J Anaesthesiol Clin Pharmacol. 2011 Jul;27(3):297-302. doi: 10.4103/0970-9185.83670. No abstract available. PMID 21897496
- [Background] Chan AK, Cheung CW, Chong YK. Alpha-2 agonists in acute pain management. Expert Opin Pharmacother. 2010 Dec;11(17):2849-68. doi: 10.1517/14656566.2010.511613. Epub 2010 Aug 13. PMID 20707597
- [Background] McQueen-Shadfar LA, Megalla SA, White WD, Olufolabi AJ, Jones CA, Habib AS. Impact of intraoperative dexmedetomidine on postoperative analgesia following gynecologic surgery. Curr Med Res Opin. 2011 Nov;27(11):2091-7. doi: 10.1185/03007995.2011.618491. Epub 2011 Sep 14. PMID 21916531
- [Background] Turgut N, Turkmen A, Gokkaya S, Altan A, Hatiboglu MA. Dexmedetomidine-based versus fentanyl-based total intravenous anesthesia for lumbar laminectomy. Minerva Anestesiol. 2008 Sep;74(9):469-74. PMID 18762754